CLINICAL TRIAL: NCT04663438
Title: First-line Atezolizumab Plus Chemotherapy in Patients With Extensive-stage Small-cell Lung Cancer:a Real World,Single Arm,Multicenter,Prospective Study in China
Brief Title: Real World Study of Efficacy and Safety of Atezolizumab Plus Chemotherapy in Chinese Patients With ES-SCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Hospital (Other Government); China-Japan Friendship Hospital (Other); Beijing Chest Hospital (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Li Zhang, Professor,Chief physician, Peking Union Medical College Hospital
Other Study IDs: ZS-2407
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: 1L ES-SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Antineoplastic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: 200/Atezolizumab combined with EC regimen Atezolizumab:1200 mg Q3w
  Interventions: Drug: Chemotherapy Drugs, Cancer
- Arm B: 100/Atezolizumab combined with chemotherapy Atezolizumab:1200mg Q3w
  Interventions: Drug: Chemotherapy Drugs, Cancer

INTERVENTIONS:
Drug: Chemotherapy Drugs, Cancer — Other chemotherapy:Irinotecan;topotecan;Enrotinib;Bevacil

SUMMARY:
The study is a prospective,multi-center,single arm,real world study to evaluate safety and performance of Atezolizumab plus chemotherapy in patients with extensive-stage small-cell lung cancer,and also to explore potential biomarkers for Immune-related Adverse Events.

DETAILED DESCRIPTION:
In 2018,the results of IMpower 133 were reported on WCLC.Meanwhile,the data was published in NEJM.Atezolizumab combined with carboplatin and etoposide for extensive stage small cell lung cancer was recommended as the first by NCCN guidelines quickly.

Atezolizumab plus chemotherapy was approved by NMPA on Feb 13,2020,making Atezolizumab for 1L ES-SCLC in China.

Real world study can reflect the efficacy and safety of treatment in clinical practice.Based on the research of public database,the prospective cohort study had been reported,but the study based on Chinese patients still left weak point.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group [VALG] staging system)
* No prior systemic treatment for ES-SCLC
* 18-80 years old, or more than 10 months of expected natural survival;
* Eastern Cooperative Oncology Group performance status of 0 or 1 or 2
* Measurable disease, as defined by RECIST v1.1 Adequate hematologic and end organ function
* Treatment-free for at least 6 months since last chemo/radiotherapy, among those treated (with curative intent) with prior chemo/radiotherapy for limited-stage SCLC
* The subject must be willing and able to participate in the study procedures and to understand and sign the informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of atezolizumab or 6 months after the final dose chemotherapy. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Patients or family members cannot understand the conditions and goals of this study.

The subject has an estimated life expectancy of less than 10 months The subject is unable or unwilling to comply with the study requirements or follow-up schedule

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is a prospective, multi-center, single-arm, real-world study to evaluate safety and performance of Atezolizumab plus chemotherapy in patients with extensive-stage small-cell lung cancer, and also to explore potential biomarkers for Immune-related Adverse Events.
  People with ES-SCLC will be included in the study according to the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
OS | Baseline until death from any cause(up to approximately 23 months)
  Duration of overall survival
irAE | Baseline until up to 90 days after end of treatment(up to approximately 46 months) and related biomarkers
  Percentage of participants with Immune-related

SECONDARY OUTCOMES:
PFS | Baseline until PD or death,whichever occurs first(up to approximately 23months)]
  Duration of Progression-Free Survival as assessed by the Investigator using Recist v1.1
Treatment related biomarkers | Baseline until PD or death,whichever occurs during this period(up to approximately 23months)]
  Biomarkers:CD 4+,CD28+,PD L1,TMB etc.
Quality of Life (QL) | Baseline until PD or death,whichever occurs during this period(up to approximately 23months)]
  QL as assessed by using EORTC
) Score | Baseline until PD or death,whichever occurs during this period(up to approximately 23months)]
  QLQ C30 Score and EORTC QLQ Lung cancer module (LC13)Score

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PhD, Principal Investigator — Peking union medical college hospital,China
Locations (1):
- Peking union medical college hospital，, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Result] Govindan R, Page N, Morgensztern D, Read W, Tierney R, Vlahiotis A, Spitznagel EL, Piccirillo J. Changing epidemiology of small-cell lung cancer in the United States over the last 30 years: analysis of the surveillance, epidemiologic, and end results database. J Clin Oncol. 2006 Oct 1;24(28):4539-44. doi: 10.1200/JCO.2005.04.4859. PMID 17008692